CLINICAL TRIAL: NCT04222959
Title: Girls Invest: A Mobile-Enabled Economic Empowerment Intervention for Girls
Brief Title: An Intervention to Reduce Risk Factors for Adolescent Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Elizabeth Reed, Principal Investigator, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21HD097496-01 (NIH)
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Behavioral Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Girls Invest Intervention (Experimental): Girls Invest intervention participants receive the app trainings and savings account with $100 deposited.
  Interventions: Behavioral: Girls Invest Intervention
- Wait-List Control Condition Participants (No Intervention): Control condition participants will be provided the Girls Invest intervention after the 6 month follow-up.

INTERVENTIONS:
Behavioral: Girls Invest Intervention — App-based trainings: The first 2 modules cover gender and cultural norms related to girls' social and economic empowerment, increasing girls' recognition of the importance of financial literacy and independence. The last 3 modules cover finance, educational loans, and employment.
  Savings account: Participants receive $100 deposited into a savings account we set up for them, conditional upon completion of app-based trainings.
  Arms: Girls Invest Intervention

SUMMARY:
Investigators will assess the preliminary effects of Girls Invest, an innovative savings intervention that aims to reduce economic, social, and health behavior risks associated with disproportionately high rates of pregnancy among US Latina adolescents. Girls Invest involves a multidisciplinary conceptual model adapting the most effective prevention strategies from the disciplines of public health and economics. Participants receive a savings account (via our collaborating bank) with $100 deposited in increments based on completion of each module of a gender and life skills training via a mobile "app."

DETAILED DESCRIPTION:
Investigators will assess the preliminary effects of Girls Invest, an innovative savings intervention that aims to reduce economic, social, and health behavior risks associated with disproportionately high rates of pregnancy among US Latina adolescents. Recommended models of adolescent pregnancy prevention in the US focus on modifying social norms (e.g., norms supporting early childbearing), as well as sexual health knowledge and skill-building; however, such efforts are not likely effective in reducing economic risk factors (e.g., financial reliance on male partners, low expectations for future career and educational achievements). Girls Invest involves a multidisciplinary conceptual model adapting the most effective prevention strategies from the disciplines of public health and economics to address social and economic risks associated with adolescent pregnancy. Participants receive a savings account (via our collaborating bank) with $100 deposited in increments based on completion of each module of a gender and life skills training via a mobile "app." Girls Invest will be evaluated among a community sample of Latina adolescents residing in economically disenfranchised neighborhoods in San Diego County with high rates of adolescent pregnancy. Adolescent pregnancy is a concern in San Diego and other US-Mexico border regions, where rates are higher compared to the rest of the US or elsewhere in Mexico. Compared to other racial/ethnic groups, Latina adolescents of Mexican origin have the highest pregnancy rates. In California, where Latinos constitute 39% of the population, 30% of all Latinas give birth prior to their 20th birthday. Latina adolescents ages 15-22 will be recruited among 18 community-based organizations and schools within low-income neighborhoods of San Diego County region. Half of the sites will be randomized to receive Girls Invest and the remaining assigned to a wait-list control condition (n= 9 sites per arm; total = 200 girls). To assess feasibility and fidelity, investigators will track (via data logs and app-based data) all aspects of recruitment, retention, and intervention completion. In-depth interviews with Girls Invest participants and focus groups with key stakeholders will inform acceptability and scalability of Girls Invest. Participants will complete a questionnaire at baseline and 6 months follow-up to assess evidence of improvements in intermediate outcomes. Regression analyses will assess treatment effects on intermediate outcomes. Investigators hypothesize that at follow-up, compared to control participants, Girls Invest participants will have reduced economic vulnerability (e.g., reduced financial reliance on male partners, improved expectations for future career and educational achievements), decreased social risks for pregnancy (e.g., intentions to delay pregnancy), and improved prioritization, knowledge of, and attitudes supportive of contraceptive use. Study findings will inform a full-scale efficacy trial of Girls Invest.

ELIGIBILITY:
Inclusion Criteria:

* age 15-22 years old
* literate in English
* have a smart phone with internet access
* have photo identification
* willing to open a savings account

Ages: 15 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

REFERENCES:
- [Background] Minnis AM, vanDommelen-Gonzalez E, Luecke E, Dow W, Bautista-Arredondo S, Padian NS. Yo Puedo--a conditional cash transfer and life skills intervention to promote adolescent sexual health: results of a randomized feasibility study in san francisco. J Adolesc Health. 2014 Jul;55(1):85-92. doi: 10.1016/j.jadohealth.2013.12.007. Epub 2014 Feb 8. PMID 24518532
- [Background] Gibbs A, Jacobson J, Kerr Wilson A. A global comprehensive review of economic interventions to prevent intimate partner violence and HIV risk behaviours. Glob Health Action. 2017 Jan-Dec;10(sup2):1290427. doi: 10.1080/16549716.2017.1290427. PMID 28467193
- [Background] Vyas S, Watts C. How does economic empowerment affect women's risk of intimate partner violence in low and middle income countries? A systematic review of published evidence. Journal of international Development. 2009;21(5):577-602.
- [Background] Jennings L, Ssewamala FM, Nabunya P. Effect of savings-led economic empowerment on HIV preventive practices among orphaned adolescents in rural Uganda: results from the Suubi-Maka randomized experiment. AIDS Care. 2016;28(3):273-82. doi: 10.1080/09540121.2015.1109585. Epub 2015 Nov 7. PMID 26548549
- [Background] Karimli L, Ssewamala FM. Do Savings Mediate Changes in Adolescents' Future Orientation and Health-Related Outcomes? Findings From Randomized Experiment in Uganda. J Adolesc Health. 2015 Oct;57(4):425-32. doi: 10.1016/j.jadohealth.2015.06.011. Epub 2015 Aug 11. PMID 26271162
- [Background] Huang J, Kim Y, Sherraden M. Material hardship and children's social-emotional development: Testing mitigating effects of Child Development Accounts in a randomized experiment. Child Care Health Dev. 2017 Jan;43(1):89-96. doi: 10.1111/cch.12385. Epub 2016 Aug 4. PMID 27488187
- [Background] Thaler, Richard, and Shlomo Benartzi. 2004. "Save More Tomorrow (TM): Using Behavioral Economics to Increase Employee Saving." Journal of Political Economy 112(S1): S164-S187.
- [Background] Schaner, S. (2017). The Persistent Power of Behavioral Change: Long-Run Impacts of Temporary Savings Subsidies for the Poor. Working paper
- [Background] Dupas P, Robinson J. Why Don't the Poor Save More? Evidence from Health Savings Experiments. Am Econ Rev. 2013 Jun;103(4):1138-71. doi: 10.1257/aer.103.4.1138. PMID 29533047
- [Background] Simons M, de Vet E, Brug J, Seidell J, Chinapaw MJ. Active and non-active video gaming among Dutch adolescents: who plays and how much? J Sci Med Sport. 2014 Nov;17(6):597-601. doi: 10.1016/j.jsams.2013.10.250. Epub 2013 Nov 9. PMID 24275124
- [Background] LeBlanc AG, Chaput JP, McFarlane A, Colley RC, Thivel D, Biddle SJ, Maddison R, Leatherdale ST, Tremblay MS. Active video games and health indicators in children and youth: a systematic review. PLoS One. 2013 Jun 14;8(6):e65351. doi: 10.1371/journal.pone.0065351. Print 2013. PMID 23799008
- [Background] Martin JA, Hamilton BE, Ventura SJ, Osterman MJ, Mathews TJ. Births: final data for 2011. Natl Vital Stat Rep. 2013 Jun 28;62(1):1-69, 72. PMID 24974591
- [Background] McDonald JA, Mojarro O, Sutton PD, Ventura SJ. Adolescent births in the border region: a descriptive analysis based on US Hispanic and Mexican birth certificates. Matern Child Health J. 2015 Jan;19(1):128-35. doi: 10.1007/s10995-014-1503-2. PMID 24820518
- [Background] Martinez G, Copen CE, Abma JC. Teenagers in the United States: sexual activity, contraceptive use, and childbearing, 2006-2010 national survey of family growth. Vital Health Stat 23. 2011 Oct;(31):1-35. PMID 22256688
- [Background] Curtin SC, Abma JC, Ventura SJ, Henshaw SK. Pregnancy rates for U.S. women continue to drop. NCHS Data Brief. 2013 Dec;(136):1-8. PMID 24314113
- [Background] Reed E, Donta B, Dasgupta A, Ghule M, Battala M, Nair S, Silverman J, Jadhav A, Palaye P, Saggurti N, Raj A. Access to Money and Relation to Women's Use of Family Planning Methods Among Young Married Women in Rural India. Matern Child Health J. 2016 Jun;20(6):1203-10. doi: 10.1007/s10995-016-1921-4. PMID 26971270
- [Background] Darney BG, Weaver MR, Sosa-Rubi SG, Walker D, Servan-Mori E, Prager S, Gakidou E. The Oportunidades conditional cash transfer program: effects on pregnancy and contraceptive use among young rural women in Mexico. Int Perspect Sex Reprod Health. 2013 Dec;39(4):205-14. doi: 10.1363/3920513. PMID 24393726
- [Background] Todd JE, Winters P, Stecklov G. Evaluating the impact of conditional cash transfer programs on fertility: the case of the Red de Protección Social in Nicaragua. Journal of Population Economics. 2012;25(1):267-290.
- [Background] Minnis AM, Marchi K, Ralph L, Biggs MA, Combellick S, Arons A, Brindis CD, Braveman P. Limited socioeconomic opportunities and Latina teen childbearing: a qualitative study of family and structural factors affecting future expectations. J Immigr Minor Health. 2013 Apr;15(2):334-40. doi: 10.1007/s10903-012-9653-z. PMID 22678305
- [Background] van Dommelen-Gonzalez E, Deardorff J, Herd D, Minnis AM. Homies with aspirations and positive peer network ties: associations with reduced frequent substance use among gang-affiliated Latino youth. J Urban Health. 2015 Apr;92(2):322-37. doi: 10.1007/s11524-014-9922-3. PMID 25649980

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: schools
Groups:
- Girls Invest Intervention: Girls Invest intervention participants were randomized by site to receive the intervention immediately upon completion of the baseline survey. Intervention participants will also complete the 6 month follow-up survey. (n=217 total participants)
  Girls Invest Mobile App Intervention: 5 levels of training on financial and health literacy Savings account and subsidies: participants receive deposits into a savings account upon completion of app-based trainings
- Wait-List Control Condition Participants: Control condition participants will be randomized upon completion of the baseline survey and put on a wait-list to receive Girls Invest behavioral intervention after the 6 month follow-up survey. (n=50 dyads; 100 total participants)
Period: Overall Study
Arm/Group | Girls Invest Intervention | Wait-List Control Condition Participants
Started | 138; 9 schools | 102; 9 schools
Completed | 62; 9 schools | 74; 9 schools
Not Completed | 76; 0 schools | 28; 0 schools
Not completed — Lost to Follow-up | 76 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Girls Invest Intervention | Wait-List Control Condition Participants | Total
Number analyzed (Participants) | 138 | 102 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 89 | 80 | 169
  Between 18 and 65 years | 49 | 22 | 71
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17 (1.5) | 17 (1.4) | 17 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 102 | 240
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: We had some participants who did not respond to this question. Thus, the total analyzed is less than the full sample.
  Participants
    number analyzed (Participants) | 118 | 88 | 206
    American Indian or Alaska Native | 10 | 5 | 15
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 0 | 0 | 0
    White | 9 | 1 | 10
    More than one race | 30 | 0 | 30
    Unknown or Not Reported | 68 | 82 | 150
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 138 | 102 | 240

OUTCOME MEASURES:

1. Primary Outcome: Sexual/Reproductive Health Behaviors
Description: Contraceptive use: Condom use and other contraception use and consistency of use.
Time Frame: 6 month follow-up
Population: Participants who reported having had sex in the past 6 months.
Measure: Count of Participants; unit: Participants
Groups:
- Girls Invest Intervention: Girls Invest intervention participants were randomized by site to receive the intervention immediately upon completion of the baseline survey.
  Girls Invest Intervention includes 2 main components:
  Girls Invest Mobile App Trainings: 5 levels of training on financial and health topics
  Savings account and subsidies: Participants receive deposits into a savings account upon completion of app-based trainings, totaling $100.
- Wait-List Control Condition Participants: Control condition participants were on a wait-list to receive Girls Invest behavioral intervention after the 6 month follow-up survey.
Arm/Group | Girls Invest Intervention | Wait-List Control Condition Participants
Number analyzed (Participants) | 55 | 39
Participants | 24 | 17

2. Primary Outcome: Financial Reliance on a Male Partner
Description: Number of participants reporting relying financially on a male partner (reported to receive spending money from a male partner or reported that a male partner buys basic necessities, such as: food, clothing, school supplies).
Time Frame: Past 6 months
Population: participants who were not lost to follow-up and responded to the item
Measure: Count of Participants; unit: Participants
Arm/Group | Girls Invest Intervention | Wait-List Control Condition Participants
Number analyzed (Participants) | 53 | 67
Participants | 11 | 12

3. Secondary Outcome: Feeling Depressed
Description: Felt down, depressed, or hopeless - 5 pt likert scale recategorized as reporting any frequency of these feelings in last 30 days versus none (assessed at 6 months follow up)
Time Frame: 6 months follow-up
Population: Participants who were not lost to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Girls Invest Intervention | Wait-List Control Condition Participants
Number analyzed (Participants) | 43 | 61
Participants | 5 | 14

4. Secondary Outcome: Felt Worried, Tense, or Anxious
Description: Felt worried, tense, or anxious - 5 pt likert scale recategorized as any frequency of these feelings in the past 30 days versus no days reporting these feelings (assessed at 6 months follow-up)
Time Frame: 6 months
Population: Participants who were not lost to follow up and responded to questions regarding feelings of depression and anxiety at follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Girls Invest Intervention | Wait-List Control Condition Participants
Number analyzed (Participants) | 43 | 61
Participants | 8 | 27

ADVERSE EVENTS:
Time Frame: We collected adverse events throughout recruitment and follow-up, spanning 1.5 years.
Groups:
- Girls Invest Intervention: Girls Invest intervention participants were randomized by site to receive the intervention immediately upon completion of the baseline survey. Intervention participants will also complete the 6 month follow-up survey. (n=217 total participants)
  Girls Invest Mobile App Intervention: App-based trainings focused on financial and health literacy. Trainings included app features such as gaming dynamics, and quizzes. Each module estimates 25 minutes to complete.
  Savings Account Subsidies: Participants receive savings deposits upon completion of the app-based trainings.
Arm/Group | Girls Invest Intervention | Wait-List Control Condition Participants
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/138 | 0/102
Other Adverse Events (participants affected / at risk) | 0/138 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT04222959/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT04222959/ICF_001.pdf